CLINICAL TRIAL: NCT02428998
Title: Safety Evaluation for 24 Weeks Intake of Korean Red Ginseng in Adults: A Randomized, Double-blind, Placebo-controlled, Parallel, Multi-center, Exploratory Trial
Brief Title: Safety for 24 Weeks Intake of Korean Red Ginseng in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Ginseng Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KGC-S-01
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Healthy; Diabetes; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Korean Red Ginseng (Experimental): Patients receive oral Korean Red Ginseng twice daily for 24 weeks. Treatment repeats every 4, 12, 24 weeks for 3 courses
  Interventions: Dietary Supplement: Korean Red Ginseng
- Placebo (Placebo Comparator): Patients receive oral placebo twice daily for 24 weeks. Treatment repeats every 4, 12,24 weeks for 3 courses
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng
  Arms: Korean Red Ginseng
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Korean Red Ginseng appears to adverse events in adults taking 24 weeks Placebo and comparative assessment. And exploratory as Korean Red Ginseng blood sugar control, reduce body fat, URTI prevention, cardiovascular risk, renal function, cholesterol, improve, fatigue, and determine the impact on biological age.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years or older
2. agree to participate in this test, voluntarily signed by the parties to a written agreement
3. In the case of women of childbearing age and confirmed negative pregnancy test, you agree to contraception during the trial period applying human characters

Exclusion Criteria:

1. Pregnant and lactating mothers
2. Patients with a history of hypersensitivity to contain ingredients that caused the test food
3. patients with severe renal disease (serum creatinine levels greater than 1.5 times if the upper limit of normal
4. Patients with severe hepatic disease, such as cirrhosis (if AST or ALT greater than three times the upper limit of normal)
5. autoimmune diseases (multiple sclerosis, lupus, rheumatoid arthritis, etc.) patients with
6. patients with uncontrolled diabetes (for HbA1c 8.0% or more)
7. Sulphonylureas, diabetic patients being treated with Insulin
8. , uncontrolled hypertension (systolic blood pressure of 150mmHg or higher or if diastolic blood pressure greater than 100mmHg)
9. uncontrolled hyperlipidemia patients (if LDL-cholesterol is 160mg / dL or higher)
10. patients with uncontrolled thyroid dysfunction
11. patients with a dementia or psychiatric problems
12. treated with systemic steroid screening visit within 1 weeks ago
13. before the screening visit 4 weeks continuously for more than two weeks, the mentally ill and insomnia patients receiving antipsychotic medication within
14. taking the medicine within 4 weeks before the screening visit
15. taking the other investigational drugs or human test food application within four weeks before the screening visit
16. taking health supplements other than vitamins and minerals within 2 weeks before randomization
17. which means in other clinical care ∙ Psychiatric Disorders diseases, cardiovascular diseases, or gastrointestinal diseases, malignant tumors such as a medical condition that is likely to affect the test result is determined to be unfit to test patient participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
All adverse events occurring up to 24 weeks time after taking the Investigational product | up to 24 weeks time after taking the Investigational product

SECONDARY OUTCOMES:
Adverse events that occurred up to 24 weeks to collect all focus point after taking the Investigational product | up to 24 weeks to collect all focus point after taking the Investigational product
Cardiovascular adverse events that occurred after taking the Investigational product | up to 24 weeks time after taking the Investigational product
Gastrointestinal adverse events that occurred after ingestion of Investigational product | up to 24 weeks time after taking the Investigational product
Neuropsychiatric adverse events that occurred after ingestion of Investigational product | up to 24 weeks time after taking the Investigational product
Grade 3 adverse events that occurred after ingestion of Investigational product | up to 24 weeks time after taking the Investigational product
Baseline by 24 weeks after the change in quality of life measures ingestion of Investigational product | up to 24 weeks time after taking the Investigational product

OTHER OUTCOMES:
glucose, insulin, HbA1c levels, HOMA-IR index variation | up to 24 weeks time after taking the Investigational product
BMI, waist circumference variation | up to 24 weeks time after taking the Investigational product
adiponectin, leptin levels of variation | up to 24 weeks time after taking the Investigational product
URTI (Upper respiratory tract infection) rates | up to 24 weeks time after taking the Investigational product
hs-CRP, IL-6, homocysteine concentration of variation | up to 24 weeks time after taking the Investigational product
eGFR, change amount of urine protein | up to 24 weeks time after taking the Investigational product
Variation of CFS (Chalder fatigue scale) | up to 24 weeks time after taking the Investigational product
variation of biological age | up to 24 weeks time after taking the Investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsoo Kim, M.D., Ph.D, Principal Investigator — The Catholic University of Korea
Locations (1):
- Catholic Universtiy of Korea. Seoul St Mary's Hospital, Seoul, South Korea